CLINICAL TRIAL: NCT00151749
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of the Efficacy and Safety of WelChol® in Type 2 Diabetes With Inadequate Glycemic Control on Insulin Therapy Alone or Insulin Therapy Combination With Other Oral Anti-diabetic Agents
Brief Title: WelChol® and Insulin in Treating Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WEL-302
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Colesevelam Hydrochloride

INTERVENTIONS:
Drug: Colesevelam hydrochloride

SUMMARY:
The purpose of the study is to see how safe and effective and tolerable the use of WelChol® is for type 2 diabetes when added to insulin alone or in combination with other anti-diabetic drugs

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 75 years, inclusive
* Diagnosed with type 2 diabetes
* Stable insulin therapy for 6 weeks
* Stable dose of any other antidiabetic medications for 90 days
* Hemoglobin A1c value between 7.5% to 9.5%
* C peptide greater than 0.5 ng/mL
* Prescribed ADA diet

Exclusion Criteria:

* History of type 1 diabetes or ketoacidosis
* History of pancreatitis
* Uncontrolled hypertension
* Allergy or toxic response to colesevelam or any of its components
* Serum LDL-C less than 60 mg/dL
* Serum TG greater than 500 mg/dL
* Body mass index (BMI) greater than 45 kg/m2-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260
Dates: Start 2004-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
- To assess the additional lowering of HbA1c achieved by
addition of WelChol® to current antidiabetic therapy

SECONDARY OUTCOMES:
To assess: the effects on fasting plasma glucose and
fructosamine; glycemic control response rate; effect on adiponectin; the effect on c-peptide; effect on c-reactive protein; effects on lipids and lipoproteins; the safety and tolerability of WelChol® as add-
on therapy to patients receiving insulin alone or with
other oral drugs

CONTACTS AND LOCATIONS:
Locations (47):
- United States (45):
  - Tuscumbia, Alabama
  - Sierra Vista, Arizona
  - Jonesboro, Arkansas
  - Searcy, Arkansas
  - Carmichael, California
  - Concord, California
  - Fullerton, California
  - La Jolla, California
  - San Diego, California
  - West Hills, California
  - Washington D.C., District of Columbia
  - Largo, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Troy, Michigan
  - Edina, Minnesota
  - Chesterfield, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Bozeman, Montana
  - Butte, Montana
  - Englewood, New Jersey
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Marion, Ohio
  - Portland, Oregon
  - Beaver, Pennsylvania
  - Charleston, South Carolina
  - Bristol, Tennessee
  - Morristown, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Midland, Texas
  - San Antonio, Texas
- Mexico City, Mexico
- Lima, Peru

REFERENCES:
- [Derived] Goldberg RB, Fonseca VA, Truitt KE, Jones MR. Efficacy and safety of colesevelam in patients with type 2 diabetes mellitus and inadequate glycemic control receiving insulin-based therapy. Arch Intern Med. 2008 Jul 28;168(14):1531-40. doi: 10.1001/archinte.168.14.1531. PMID 18663165